CLINICAL TRIAL: NCT03554356
Title: Nitrous Oxide For Endoscopic Ablation of Refractory Barrett's Esophagus (NO FEAR-BE)
Acronym: NO FEAR-BE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: PENTAX of America, Inc. (Unknown); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0388
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Intestinal Metaplasia; Esophageal Dysplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cryoballoon Focal Ablation System (CbFAS) Treatment (Experimental): Subjects undergoing CbFAS treatment as part of their clinical care for their condition.
  Interventions: Device: CryoBalloon Focal Ablation System

INTERVENTIONS:
Device: CryoBalloon Focal Ablation System — CryoBalloon Focal Ablation System

SUMMARY:
A multicenter, prospective, single arm, non randomized clinical trial to evaluate the safety and efficacy of the C2 CryoBalloon Focal Ablation System (CbFAS) for the treatment of persistent dysplasia or intestinal metaplasia (IM) in the tubular esophagus after 3 or more radiofrequency ablations (RFA) for dysplastic BE, or <50% eradication of Barrett's Esophagus (BE) after 2 RFA treatments.

DETAILED DESCRIPTION:
Eligibility will be determined based on historical local pathology and medical record information. Informed consent will be obtained and eligible subjects will be treated with the Cryoballoon Focal Ablation System (CbFAS) at baseline.

Subjects will return every 3 months +/- 6 weeks for repeat treatment for up to 12 months OR until complete eradication of intestinal metaplasia (CEIM) and complete eradication of dysplasia (CED) are achieved (at which point subjects enter the follow-up phase), whichever occurs first.

Treatment procedures will be performed on an outpatient basis according to the site's standards of care for anesthesia and sedation during esophagogastroduodenoscopy (EGD) procedures. EGD examinations will be performed using high definition White Light Endoscopy (WLE), plus Narrow Band Imaging (NBI) or i-SCAN to assess BE measurements and identify tissue landmarks and ablation zones.

A high definition endoscope will be used for all ablations performed with the CryoBalloon Focal Ablation System (CbFAS). The System will be used according to the instructions for use provided with the product and in accordance with the current standard of care for treatment of BE.

Repeat cryoablation may be performed if esophageal columnar mucosa is visible on EGD or if intervening biopsies (if a site chooses to obtain intervening biopsies as standard of care) are positive for any esophageal columnar epithelium until complete eradication of all unwanted tissue is achieved.

Intervening endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) after enrollment may be performed for nodular areas detected after baseline. EMR/ESD may be performed at the same session as the cryoablation if the EMR/ESD site is >=3cm away from the ablation target site. Cryoablation should be performed before EMR/ESD. If the EMR/ESD site is within 3cm of target treatment area, then CbFAS will be delayed for at least 6 weeks.

Residual islands of columnar mucosa of <5 mm in diameter each and <= 3 total can be treated with Argon Plasma Coagulation (APC) and/or CbFAS at the discretion of the treating physician to avoid over treatment of neo-squamous mucosa.

Stenosis requiring treatment based on the physician's discretion, which develops after enrollment, will be treated with standard of care balloon- or wire-guided dilation. Cryoablation may be performed at the same session if the dilated site is >= 3 cm from the target cryoablation site. Otherwise, cryoablation will be postponed to another visit within 1 month +/- 2 weeks.

When CbFAS treatment is received, subjects will be asked to complete assessments immediately after CbFAS treatment, and will be contacted 1 day, 7 days, and 30 days after the procedure.

If no visible BE is present during the endoscopy, then at least eight (8) biopsies in total will be obtained: at least four (4) from the distal esophagus in the neosquamous epithelium and at least four (4 from the gastroesophageal junction (GEJ), top of gastric folds (TGF), or gastric cardia. Additional biopsies may be taken as per standard of care guidelines at the site.

Biopsies will be read by local expert pathologist. If biopsies indicate CEIM and CED, then subjects will enter the 12 month follow-up phase. If biopsies do not indicate CEIM and CED, then subjects will return for additional CbFAS treatment in 3 months +/-6 weeks.

Non-responders are defined as subjects who have not achieved CEIM and CED at 12 months post baseline CbFAS treatment. Non-responders at 12 months will exit the study and continue treatment at the physician's discretion and according to standard of care at each site.

Subjects who achieve CEIM and CED within 12 months of the baseline CbFAS procedure will enter a 12 month follow-up phase. Subjects will be followed per routine care guidelines for their condition, described below:

Subjects with baseline LGD will return at 6 and 12 months from the initial CEIM and CED date for follow-up (+/-4 weeks). Subjects with baseline HGD or IMC will return at 3, 6, 9, and 12 months from initial CEIM and CED date for follow-up (+/- 4 weeks).

During follow-up procedures, high definition WLE, plus NBI or i-SCAN will be used to assess BE measurements, and then at least eight (8) biopsies in total will be obtained: at least four (4) from the distal esophagus in the neosquamous epithelium and at least four (4 from the gastroesophageal junction (GEJ), top of gastric folds (TGF), or gastric cardia. Additional biopsies may be taken as per standard of care guidelines at the site. Biopsies will be read by local expert pathologist.

If recurrent BE is detected during follow-up endoscopy with biopsy demonstrating compatible histology, then subjects will be exited from the study and treated at the physician's discretion.

Study participation is complete if: 1) Subject has not reached CEIM and CED at 12 month post baseline treatment; or 2) If BE or dysplasia recur after initial CEIM and CED post enrollment; 3) Subject is discovered to be ineligible after enrollment; or 4) After completion of the 12 month follow-up EGD with biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. History of BE with LGD or HGD confirmed with biopsy, or resected intramucosal cancer (IMC) with low risk of recurrence defined as EMR/ESD pathology results negative for: positive margin, >T1a stage, poorly differentiated carcinoma, and lymphovascular invasion.
2. Prior treatment with RFA who meet either of the following criteria at the enrolling EGD:

   2.1. History of at least 3 RFA treatments, with one or more of the following:
   * 2.1.1. Residual BE Prague >=C1
   * 2.1.2. Residual BE >=M1
   * 2.1.3. One or more islands of residual BE >=1 cm in diameter
   * 2.1.4. Any residual dysplasia in tubular esophagus 2.2. History of at least 2 RFA treatments and < 50% eradication of BE, as judged by estimation of the treating physician.
3. 18 or older years of age at time of consent.
4. Provides written informed consent.
5. Willing to undergo an alternative approved standard of care treatment for their condition.
6. Willing and able to comply with study requirements for follow-up.
7. No prior history of balloon or spray cryotherapy esophageal treatment. Prior APC is allowable.

Exclusion Criteria:

1. Residual BE Prague length measuring >C3 or >M8 after RFA treatment.
2. Dysplasia or IM confined only to the gastric cardia.
3. Pre-existing esophageal stenosis/stricture preventing advancement of a therapeutic endoscope during screening/baseline EGD. Subjects are eligible if the stenosis/stricture is dilated to at least 15mm, but baseline treatment may need to be delayed per protocol.
4. Symptomatic, untreated esophageal strictures.
5. 5. Any endoscopically visualized abnormalities such as ulcers, masses, or nodules found in the BE during screening/baseline EGD. Subjects with nodular dysplasia or IMC identified during screening/baseline EGD may be treated with EMR or ESD and return for baseline treatment in this study at least 6 weeks later given that: 5.1. Follow-up endoscopy must be negative for nodular dysplasia (visually clear of nodular dysplasia).

   5.2. Patients with IMC must be at low risk for recurrence, confirmed by EMR/ESD pathology results negative for: positive margin, >T1a stage, poorly differentiated carcinoma, and lymphovascular invasion.
6. EMR or ESD < 6 weeks prior to baseline treatment.
7. Untreated invasive esophageal malignancy, including margin-positive EMR/ESD.
8. Active reflux esophagitis grade B or higher in the BE assessed during screening/baseline EGD.
9. Severe medical comorbidities precluding endoscopy or limiting life expectancy to less than 2 years in the judgment of the endoscopist.
10. Uncontrolled coagulopathy.
11. Inability to hold use of anti-coagulation medications or non-aspirin anti-platelet agents (APAs) for the duration recommended per ASGE guidelines for a high-risk endoscopy procedure.
12. Active fungal esophagitis.
13. Known portal hypertension, visible esophageal varices, or history of esophageal varices.
14. General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation.
15. Pregnant or planning to become pregnant during period of study participation.
16. Patient refuses or is unable to provide written informed consent.
17. Prior esophageal surgery with the exception of uncomplicated nissen fundoplication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of all treated Subjects with complete eradication of all intestinal metaplasia (CEIM) within 12 months of enrollment. | 12 months
Percentage of all treated subjects with complete eradication of dysplasia (CED) within 12 months of enrollment | 12 months
  Stratified by prior type of ablation treatment and baseline grade (LGD or HGD) will also be reported.
Incidence of CryoBalloon-related serious adverse events | 12 months
  Relation of serious adverse events to CryoBalloon device will be assessed by the PI

SECONDARY OUTCOMES:
Technical success rate | At end of treatment period, up to 12 months
  The device worked as expected on every application, defined as proportion of all CbFAS that perform as intended.
Procedure success rate | At end of treatment period, up to 12 months
  All columnar tissue that was planned to be treated was treated.
Progression rate | At end of treatment period, up to 12 months
  Percentage of subjects with progression of dysplasia from LGD to HGD or esophageal cancer, or progression of HGD to cancer at 12 months from enrollment date.
Survival curve analysis - time to CEIM | At end of treatment period, up to 12 months
  Time to complete eradication of intestinal metaplasia (CEIM). Survival curve analysis from first treatment.
Survival curve analysis - time to progression | At end of treatment period, up to 12 months
  Time to progression of dysplasia from LGD to HGD or esophageal cancer, or progression of HGD to cancer at 12 months from enrollment date. Survival curve analysis from first treatment.
Survival curve analysis - time to recurrence | At end of treatment period, up to 12 months
  Time to recurrence. Survival curve analysis from first treatment.
Risk factors associated with failure to respond to CryoBalloon ablation | At end of treatment period, up to 12 months
  Risk factors associated with failure to respond to CryoBalloon ablation
Median number of CryoBalloon ablation treatments required to achieve CED and CEIM by 12 months from enrollment date. | At end of treatment period, up to 12 months
  Median number of CryoBalloon ablation treatments required to achieve CED and CEIM by 12 months from enrollment date.
Mean number of CryoBalloon ablation treatments required to achieve CED and CEIM by 12 months from enrollment date. | At end of treatment period, up to 12 months
  Mean number of CryoBalloon ablation treatments required to achieve CED and CEIM by 12 months from enrollment date.
Proportion of subjects requiring narcotic analgesic - Day 1 | Day 1
  Proportion of subjects requiring narcotic analgesic at day 1 post treatment.
Proportion of subjects requiring narcotic analgesic - Day 7 | Day 7
  Proportion of subjects requiring narcotic analgesic at day 7 post treatment.
Proportion of subjects requiring narcotic analgesic - Day 30 | Day 30
  Proportion of subjects requiring narcotic analgesic at day 30 post treatment.
Median pain score - Day 1 | Day 1
  Median pain score immediately post-procedure day 1 as assessed by self-reported pain scale (0-10) where 0 is no pain and 10 is worst pain imaginable. Higher scores indicate more severe pain.
Median pain score - Day 7 | Day 7
  Median pain score 7 days after treatment as assessed by self-reported pain scale (0-10) where 0 is no pain and 10 is worst pain imaginable. Higher scores indicate more severe pain.
Median pain score - Day 30 | Day 30
  Median pain score 30 days after treatment as assessed by self-reported pain scale (0-10) where 0 is no pain and 10 is worst pain imaginable. Higher scores indicate more severe pain.
Mean pain score - Day 1 | Day 1
  Mean pain score immediately post-procedure day 1 as assessed by self-reported pain scale (0-10) where 0 is no pain and 10 is worst pain imaginable. Higher scores indicate more severe pain.
Mean pain score - Day 7 | Day 7
  Mean pain score 7 days after treatment as assessed by self-reported pain scale (0-10) where 0 is no pain and 10 is worst pain imaginable. Higher scores indicate more severe pain.
Mean pain score - Day 30 | Day 30
  Mean pain score 30 days after treatment as assessed by self-reported pain scale (0-10) where 0 is no pain and 10 is worst pain imaginable. Higher scores indicate more severe pain.
Proportion of Barrett's Esophagus surface area reverted to neosquamous epithelium | At end of treatment period, up to 12 months
  For those who do not achieve CEIM and CED at 12 months from enrollment date, proportion of Barrett's Esophagus surface area reverted to neosquamous epithelium based on physician report.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Shaheeen, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Northwell Health, Lake Success, New York
  - Columbia University, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UTHealth Science Center/Herman Memorial, Houston, Texas